CONSENT Exempt

Protocol Number: 2023E0915 Approval date: 9/29/23

Version: 1

1 2

# The Ohio State University Consent to Participate in Research

3 4

Study Title: Stop Addiction Stigma

Researcher: Gretchen McNally, PhD, ANP-BC, AOCNP

Sponsor: None

5 6 7

This is a consent form for research participation. It contains important information about this study and what to expect if you decide to participate.

8 9

10

## Your participation is voluntary.

- Please consider the information carefully. Feel free to ask questions before making your 11
- decision whether or not to participate. If you decide to participate, you will be asked to sign 12
- this form and will receive a copy of the form. 13

14 15

16

17

**Purpose:** The purpose of the study is to collect data to gather information on how language may influence beliefs. Your responses will help us gather information that will help develop future educational programs and research, with the ultimate goal of improving care and outcomes of our patients.

18 19

20 21

22

23

24

25

**Procedures/Tasks:** The survey will be distributed via email to OSUWMC department of rehabilitation services personnel. This includes physical therapy, occupational therapy, speech therapy, recreational therapy, and administrative personnel. Rehabilitation services include over 700 employees, operating within the OSUWMC hospitals and inpatient units, as well at satellite and ambulatory sites across central Ohio. It is estimated that 150-200 personnel will attend the live SAS session.

26 27

28 29

**Duration:** There will be 3 surveys in total. The surveys will be collected before the Lunch and Learn, immediately after the Lunch and Learn, and then 8 weeks later.

30 31

CONSENT Pro

Protocol Number: 2023E0915

Approval date: 9/29/23

Version: 1

You may leave the study at any time. If you decide to stop participating in the study, there will be no penalty to you, and you will not lose any benefits to which you are otherwise entitled. Your decision will not affect your future relationship with The Ohio State University.

**Risks and Benefits:** Risks to participants may involve the stress and discomfort associated with the sharing of beliefs related to individuals with substance use. This is thought to be a possible, though unlikely, risk to participants.

## **Confidentiality:**

We will work to make sure that no one sees your online responses without approval. However, because we are using the Internet, there is a chance that someone could access your online responses without permission. In some cases, this information could be used to identify you.

Efforts will be made to keep your study-related information confidential. However, there may be circumstances where this information must be released. For example, personal information regarding your participation in this study may be disclosed if required by state law. Also, your records may be reviewed by the following groups (as applicable to the research):

Office for Human Research Protections or other federal, state, or international regulatory agencies;
 The Ohio State University Institutional Review Board or Office of Responsible

 Research Practices;

• Authorized Ohio State University staff not involved in the study may be aware that

• The sponsor, if any, or agency (including the Food and Drug Administration for FDA-regulated research) supporting the study.

you are participating in a research study and have access to your information; and

Future Research: Your de-identified information may be used or shared with other researchers without your additional informed consent.

#### **Incentives:**

Participants will receive a certificate for a \$5 Amazon gift card via email once each survey is completed, even if incomplete (i.e. questions were skipped). By law, payments to participants are considered taxable income.

## **Participant Rights:**

 CONSENT Protocol Number:
Exempt Approval date:

Approval date: 9/29/23
Version: 1

You may refuse to participate in this study without penalty or loss of benefits to which you are otherwise entitled. If you are a student or employee at Ohio State, your decision will not affect your grades or employment status.

78 79

80

If you choose to participate in the study, you may discontinue participation at any time without penalty or loss of benefits. By signing this form, you do not give up any personal legal rights you may have as a participant in this study.

818283

This study has been determined Exempt from IRB review.

84 85

## **Contacts and Questions:**

86

- For questions, concerns or complaints about the study, or if you feel you have been harmed as a result of study participation, you may contact:
- 69 Gretchen A. McNally, PhD, ANP-BC, AOCNP at 614-293-3196.
- 90 For questions about your rights as a participant in this study or to discuss other study-related
- oncerns or complaints with someone who is not part of the research team, you may contact
- 92 the Office of Responsible Research Practices at 1-800-678-6251 or hsconcerns@osu.edu.

93

# **Providing Consent**

94 95 96

97 98 I have read (or someone has read to me) this page and I am aware that I am being asked to participate in a research study. I have had the opportunity to ask questions and have had them answered to my satisfaction. I voluntarily agree to participate in this study. I am not giving up any legal rights by agreeing to participate.

99 100 101

To print or save a copy of this page, select the print button on your web browser.

102103

104

Please click the button below to proceed and participate in this study. If you do not wish to participate, please close out your browser window.